CLINICAL TRIAL: NCT01697605
Title: A Phase I Study of Oral BGJ398 in Asian Patients With Advanced Solid Tumor Having Alterations of the FGF-R Pathway
Brief Title: A Phase I Study of Oral BGJ398 in Asian Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBGJ398X1101
Record Dates: First submitted 2012-09-19; First posted 2012-10-02 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-03

CONDITIONS: Tumor With Alterations of the FGF-R
Keywords: Phase I, open-label, dose escalation, BGJ398, Japanese, Asian, FGF-R
MeSH Terms: interventions — infigratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BGJ398 (Experimental): Eligible participants received oral BGJ398 once daily or twice daily. Patients may continue treatment with BGJ398 until the patient experiences unacceptable toxicity or progressive disease.
  Interventions: Drug: BGJ398

INTERVENTIONS:
Drug: BGJ398

SUMMARY:
This study will evaluate safety and tolerability to determine the Maximum tolerated dose (MTD) and/or Recommended dose (RD).

DETAILED DESCRIPTION:
This is a multi-center, open label, dose finding, phase I study of oral single agent BGJ398, administered on a continuous once and/or twice daily schedule.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced solid tumors with FGF-R alteration
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate organ function

Exclusion Criteria:

* Patients with untreated and/or symptomatic metastatic Central Nerve System (CNS) disease
* Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-10-19 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Incidence rate and category of dose limiting toxicities (DLTs) | First cycle of 28 days
  Maximum tolerated dose (MTD) and/or Recommended dose (RD) of single agent oral BGJ398

SECONDARY OUTCOMES:
Frequency of all Adverse Events (AEs) and Serious Advers Events (SAEs) | From within 21 days of first treatment to 28 days after treatment discontinuation
  To characterize the safety and tolerability of oral BGJ398
Changes in hematology and chemistry values | From baseline to 28 days after treatment discontinuation
  hematology and chemistry values
Assessments of physical examinations, vital signs and electrocardiograms (ECGs) | Participants will be followed for the duration of treatment, an expected average of 24 weeks.
Time vs. concentration profiles | 1 to 10 time points (0, 0.25, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose) up to 24 weeks
  To determine the pharmacokinetic (PK) profiles (Cmax, AUC, Tmax, T1/2, etc) of oral BGJ398 including known pharmacologically active metabolites
Preliminary anti-tumor activity | Participants will be followed for the duration of treatment, an expected average of 24 weeks.
  Assessed based on RECIST version 1.1
Best overall response (BOR) | Participants will be followed for the duration of treatment, an expected average of 24 weeks.
  Assessed by investigator per RECIST version 1.1. BOR is the best response recorded until disease progression.
Overall response rate (ORR) | Participants will be followed for the duration of treatment, an expected average of 24 weeks.
  Assessed by investigator per RECIST version 1.1. ORR is the proportion of patients with a best overall response of Complete Response (CR) or Partial Response (PR).
Progression-free survival (PFS) | From date of end of treatment until the date of progression, or date of death, or starting date of a new anticancer therapy, assessed up to 100 months.
  PFS is defined as the times from the date of first dose of BGJ398 to the date of the first documented disease progression, date of death due to any cause or until a new anticancer therapy is initiated, whichever occurs first.
Duration of all Adverse Events (AEs) | From within 21 days of first treatment to 28 days after treatment discontinuation
  To characterize the safety and tolerability of oral BGJ398
Duration of Serious Advers Events (SAEs) | From within 21 days of first treatment to 28 days after treatment discontinuation
  To characterize the safety and tolerability of oral BGJ398
Severity of all Adverse Events (AEs) | From within 21 days of first treatment to 28 days after treatment discontinuation
  To characterize the safety and tolerability of oral BGJ398
Severity of all Serious Advers Events (SAEs) | From within 21 days of first treatment to 28 days after treatment discontinuation
  To characterize the safety and tolerability of oral BGJ398

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- China (3):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Guangzhou
- Japan (5):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East (NCEE), Kashiwa, Chiba
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Sayama, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CBGJ398X1101 can be found on the Novartis Clinical Trials Results website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17561